CLINICAL TRIAL: NCT06321042
Title: Evaluation of the Clinical Outcomes of the Total Knee Prosthesis With Posterior Stabilization Implanted With the Use of Inertial Sensors
Brief Title: Evaluation of the Clinical Outcomes of the Total Knee ps Prosthesis Implanted With the Use of Inertial Sensors
Acronym: SYMPHO-EM
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: SYMPHO-EM
Record Dates: First submitted 2024-01-13; First posted 2024-03-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-03

CONDITIONS: Prosthesis Durability
MeSH Terms: conditions — Prosthesis Failure | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient treated with PS Link Symphoknee prosthesis and Orthokey perseus alignment device
  Interventions: Device: Knee arthroplasty

INTERVENTIONS:
Device: Knee arthroplasty — Knee arthroplasty surgery with perseus orthokey alignment device

SUMMARY:
evaluate the clinical outcome of the implantation of a specific primary TKA model implanted with the aid of inertial sensors for the execution of bone cuts through the administration of questionnaires for the calculation of clinical-functional scores;

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 50 years of age or older and less than 85 years of age (>50 and <85 years) who are candidates for primary cemented total knee replacement based on physical examination and medical history, including diagnosis of severe knee pain and disability due to at least one of the following causes:

   * to. Primary or secondary osteoarthritis
   * b. Collagen disorders and/or avascular necrosis of femoral condyle
   * c. Moderate valgus, varus or flexion deformities (HKA between ± 10°, flexion contracture <10°) -
2. Patients consent and able to complete scheduled study procedures and follow-up assessments.
3. Patients informed about the nature of the study who signed the "informed consent" approved by the ethics committee.

Exclusion Criteria:

* Simultaneous participation in other studies
* Patients not capable of understanding and wanting and therefore unable to sign the informed consent
* Patients who have already undergone hip or ankle arthroplasty, previous osteotomy, with severe axial deformities or suffering from rheumatoid arthritis, diabetes or neuromuscular diseases.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients candidates to TKA surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score | at baseline (day 0)
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Knee Society Score | 6 months
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Knee Society Score | 12 months
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Knee Society Score | 24 months
  Two sections, one evaluating the patient's function and one for his clinical conditions, overall score goes from 0 to 100
Western Ontario and McMaster Universities Arthritis Index | at baseline (day 0)
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Western Ontario and McMaster Universities Arthritis Index | 6 months
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Western Ontario and McMaster Universities Arthritis Index | 12 months
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Western Ontario and McMaster Universities Arthritis Index | 24 months
  The test evaluates main aspects of arthritis such as pain, stiffness articulation and functionality. The score goes from 0 to 96
Knee injury and Osteoarthritis Outcome Score | at baseline (day 0)
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). the score goes from 0 to 100
Knee injury and Osteoarthritis Outcome Score | 6 months
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). the score goes from 0 to 100
Knee injury and Osteoarthritis Outcome Score | 12 months
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). the score goes from 0 to 100
Knee injury and Osteoarthritis Outcome Score | 24 months
  The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL). the score goes from 0 to 100
36-Item Short Form Health Survey | at baseline (day 0)
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.
36-Item Short Form Health Survey | 6 months
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.
36-Item Short Form Health Survey | 12 months
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.
36-Item Short Form Health Survey | 24 months
  is a valid and reliable tool for measuring health outcomes in patients with musculoskeletal pain, but its sensitivity to clinical changes in patients with specific disorders may be limited, rated on a scale of 0 to 100, with 0 and 100 being minimum and maximum possible scores.
Forgotten joint score | at baseline (day 0)
  a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint
Forgotten joint score | 6 months
  a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint
Forgotten joint score | 12 months
  a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint
Forgotten joint score | 24 months
  a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint

SECONDARY OUTCOMES:
Radiographic evaluation of prosthetic femoral component positioning | 5 days after index surgery
  measurement of prosthetic femoral component alignment according to femoral mechanical axis

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Zaffagnini, Bologna, Italia, Italy